CLINICAL TRIAL: NCT05168007
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multi-Center, Fixed-Dose, Phase 3 Clinical Trial Evaluating the Efficacy and Safety of WID-RGC20 3 mg/Day and 6 mg/Day in Patients With Acute Psychotic Episode of Schizophrenia
Brief Title: Study Evaluating the Efficacy and Safety of WID-RGC20(Cariprazine) in Patients With Schizophrenia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Whanin Pharmaceutical Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WID-RGC20-P3
Record Dates: First submitted 2021-11-26; First posted 2021-12-22 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cariprazine 3mg/day (Experimental): WID-RGC20(Cariprazine) 3 mg/day
  Interventions: Drug: WID-RGC20(Cariprazine) 3mg/day
- Cariprazine 6mg/day (Experimental): WID-RGC20(Cariprazine) 6 mg/day
  Interventions: Drug: WID-RGC20(Cariprazine) 6mg/day
- Placebo (Placebo Comparator): Placebo for WID-RGC20(Cariprazine) 3 mg/day or 6mg/day
  Interventions: Drug: Placebo for WID-RGC20(Cariprazine) 3mg/day or 6mg/day

INTERVENTIONS:
Drug: WID-RGC20(Cariprazine) 3mg/day — The initial dose is WID-RGC20(Cariprazine) 1.5mg/day, followed by an up-titration of 1.5mg/day until the target dose(3mg/day) is achieved. The investigational product is administered during the double-blind treatment period(6 weeks).
  Arms: Cariprazine 3mg/day
Drug: WID-RGC20(Cariprazine) 6mg/day — The initial dose is WID-RGC20(Cariprazine) 1.5mg/day, followed by an up-titration of 1.5mg/day until the target dose(6mg/day) is achieved. The investigational product is administered during the double-blind treatment period(6 weeks).
  Arms: Cariprazine 6mg/day
Drug: Placebo for WID-RGC20(Cariprazine) 3mg/day or 6mg/day — The placebo comparator is administered during the double-blind treatment period(6 weeks).
  Arms: Placebo

SUMMARY:
This Study is a Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multi-Center, Fixed-Dose, Phase 3 Clinical Trial Evaluating the Efficacy and Safety of WID-RGC20 3 mg/day and 6 mg/day in Patients with Acute Psychotic Episode of Schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 19 ≤ age < 65 years
* At least 1 year of schizophrenia diagnosed according to DSM-5 criteria(295.90)
* At least 1 psychotic episode within 1 year
* Current psychotic episode(acute exacerbation of schizophrenia) within 2 weeks
* 80 ≤ PANSS total score ≤ 120
* Rating of at least 4(moderate) on at least 2 of the following 4 PANSS positive symptoms
* CGI-S score ≥ 4
* Patients who can be hospitalized during the screening period and at least 3 weeks of the initial double-blind treatment phase

Exclusion Criteria:

1. Psychiatric Criteria

   * Medical history except schizophrenia specified in protocol
   * First-episode psychosis
   * Treatment-resistant schizophrenia within 2 years
   * Positive result from the blood alcohol concentration(BAC) test or the urine drug screen(UDS)
   * Have suicide risk
2. Treatment-related Criteria

   * Electroconvulsive therapy(ECT) within 12 weeks or Previous lack of response to ECT
   * Concomitant treatment with 3 or more antipsychotics within 12 weeks
   * Treatment with flunitrazepam or LAI antipsychotics less than 1 cycle or clozapine within 24 weeks
   * Treatment with CYP3A4 inducers or potent CYP3A4 inhibitors
   * Treatment with amiodarone or systemic corticosteroids for ≥ 12 weeks within 1 year
   * Required prohibited concomitant medication during the study period
   * Prior participation in any clinical trials of Cariprazine
3. Other

   * Ophthalmic medical findings or related history(ex. uncontrolled diabetes or hypertension)
   * Abnormal laboratory findings specified in protocol
   * Not suitable for any other reason, as judged by the investigator

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 342 (Estimated)
Dates: Start 2021-11-19 (Actual); Primary Completion 2023-07-17 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Positive And Negative Syndrome Scale(PANSS) total score | at Week 6
  Change from baseline in Positive And Negative Syndrome Scale(PANSS) total score at Week 6

SECONDARY OUTCOMES:
Clinical Global Impressions-Severity(CGI-S) | at Week 6
  Change from baseline in Clinical Global Impressions-Severity(CGI-S) at Week 6

OTHER OUTCOMES:
Positive And Negative Syndrome Scale(PANSS) total score | up to 5 weeks
  Change from baseline in Positive And Negative Syndrome Scale(PANSS) total score at Week 1, 2, 3, 4, 5
Clinical Global Impressions-Severity(CGI-S) | up to 5 weeks
  Change from baseline in Clinical Global Impressions-Severity(CGI-S) at Week 1, 2, 3, 4, 5
Clinical Global Impressions-Improvement(CGI-I) | up to 6 weeks
  Clinical Global Impressions-Improvement(CGI-I) at Week 1, 2, 3, 4, 5, 6
Positive And Negative Syndrome Scale(PANSS) positive score | up to 6 weeks
  Change from baseline in Positive And Negative Syndrome Scale(PANSS) positive score by Week 6
Positive And Negative Syndrome Scale(PANSS) negative score | up to 6 weeks
  Change from baseline in Positive And Negative Syndrome Scale(PANSS) negative score by Week 6
Positive And Negative Syndrome Scale(PANSS) responder | at Week 6
  Percentage of subjects with at least 30% reduction in the Positive And Negative Syndrome Scale(PANSS) total score at Week 6 compared with baseline
Adverse event(AE) | up to 8 weeks
  Incidence of Adverse event(AE)s by Week 8
Suicidal ideation and behavior | up to 8 weeks
  Incidence of suicidal ideation and behavior by Week 8
Extrapyramidal Symptoms(EPS) | up to 6 weeks
  Incidence of Extrapyramidal Symptoms(EPS) by Week 6
Laboratory test | up to 6 weeks
  Change from baseline in clinical laboratory tests by Week 6

CONTACTS AND LOCATIONS:
Locations (1):
- Whan In Pharm., Seoul, South Korea